CLINICAL TRIAL: NCT02438540
Title: Placebo-controlled, Randomized, Double Blind Trial, What is the Therapeutic Effect of Metformin and Acupuncture Combined Therapy in Comparison With Metformin Monotherapy on Weight Loss and Insulin Sensitivity in Diabetic Patients
Brief Title: Comparative the Effect of Metformin and Acupuncture on Weight Loss and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amir Firouzjaei (Other)
Responsible Party: Sponsor-Investigator, Amir Firouzjaei, Clinical PhD in Chinese medicine, Nanjing University of Traditional Chinese Medicine
Organization: Nanjing University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NanjingUTCM
Record Dates: First submitted 2015-04-21; First posted 2015-05-08 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Insulin Sensitivity; Obesity
Keywords: acupuncture; obesity; type 2 diabetic mellitus; insulin sensitivity; metformin; inflammatory factor; adipokines; lipid profile
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Metformin; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin & acupuncture (Experimental): Metformin 500 mg (one/two/three times per day), to control their diabetes during the period of this study as previously, and acupuncture treatment including electro body acupuncture and Auricular acupuncture for 30 minutes, 10 times, every other day, for 3 weeks.
  Interventions: Drug: metformin; Other: acupuncture
- metformin & placebo (Placebo Comparator): Metformin 500 mg (one/two/three times per day), to control their diabetes during the period of this study as previously, and placebo acupuncture treatment, needling not in right acupoints and EA machine was switched off during 30 minutes of therapeutic time. For ear acupuncture was just used sticky layers without seeds. All placebo treatment used for 30 minutes, 10 times, every other day, for 3 weeks.
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin — metformin tablet 500 mg
Other: acupuncture — Electro body acupuncture and auricular acupuncture
  Arms: metformin & acupuncture

SUMMARY:
The investigators designed this randomized double blind (patients/ assessor) clinical trial to compare the therapeutic effects of Metformin monotherapy with Metformin and acupuncture combined therapy on weight loss and insulin sensitivity among overweight/obese type 2 diabetes mellitus (T2DM) patients. We compared the inflammatory markers, lipid profiles, and adipokines in overweight/obese T2DM patients receiving the combined therapy to those receiving the Metformin monotherapy, to understand whether acupuncture plus Metformin is a better approach then Metformin only on treating diabetes.

DETAILED DESCRIPTION:
From 39 participants, 19 participants were sent to case group and 20 to control group according to above mentioned method of randomization by independent research assistant. In the case group enrolled participants were treated with Metformin monotherapy and received electro acupuncture (EA) and Auricular acupuncture at the selected acupoints, and participants in a control group were treated with Metformin monotherapy and received sham EA. All patients were blinded to treatment assignment during the period of study and assessor was blinded to name of the patients and results as well. IR was calculated by the homeostasis model assessment of insulin resistance (HOMA-IR) proposed by Matthews et al. HOMA-IR = (fasting insulin (mmol/L) × fasting glucose (µIU/ml))/22.5; body height was measured to an accuracy of +/-0.1cm; body weight was measured while the subjects were dressed in light clothing after an overnight fasting by standard scale to an accuracy of +/-0.1 kg; The body mass index (BMI) was calculated by dividing weight (kg) into height (squared m²). Blood markers including fasting blood sugar (FBS), fasting insulin (FINS), interleukin-6 (IL-6), tumor necrosis α (TNFα), C reactive protein (CRP), leptin, adiponectin, resistin, glucagon-like peptide-1 (GLP-1), HOMA index , free fatty acid (FFAs), low density lipoprotein cholesterol (LDLc), high density lipoprotein cholesterol (HDLc) , and ceramides; were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient after 8 hours overnight fasting, before treatment, and for FBS, FINS and HOMA index 30 min after treatment additionally, 3 times during the study (in the beginning, in the 5th time and at the end) from both groups, with the chosen for this research standard range. All data with standard range were managed by Epi-data software, then analyzed by Statistical Package for the Social Sciences (SPSS) software 15.0.0 (6 Sep 2006). The investigators statistics method included T-test and repeated measures ANOVA. P-Value<0.05 was statistically significant in this trial

ELIGIBILITY:
Inclusion Criteria:

* Who had been diagnosed with type 2 diabetes mellitus and has using Metformin monotherapy as well to control their diabetes during the period of this study as previously (500 mg one/two/three times per day)
* All patients were overweight according to BMI ≥25

Exclusion Criteria:

* Individuals with nephritic syndrome (urine protein over 3.5 g/day), edema or renal failure (serum creatinine over 115 µmol/L)
* Individuals who had been diagnosed with heart failure (NYHA Fc III-IV) or who had been a pacemaker implanted
* Individuals with abnormal liver dysfunction (GOT and glutamate-pyruvate transaminase (GPT) levels twofold above the normal range) or a diagnosis of liver cirrhosis
* Individuals with a high HbA1C level (HbA1C above 9 %)
* Pregnant women
* Individuals who were receiving insulin therapy already
* Individuals who receive other therapy or had any change at dosage during the period of therapy
* Individuals who were suffering from endocrine abnormalities such as Thyroid disease, polycystic ovary syndrome (PCOS), etc
* Individuals who were receiving weight loss medicine, anti depressant agents' or hormonal medicines during the last 3 months and the period of study
* Individuals who were suffering from a homeostasis disorder or other systemic disease
* Individuals who did not comply(signed informed consent) with the treatment during the study period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Firouzjaei, Clinical PhD, Principal Investigator — Nanjing University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 participants took part in trial. 4 of them were excluded from the trial according to including and excluding criteria. At last, 39 participants were distributed by permuted-block randomization.
Groups:
- Metformin & Acupuncture: Metformin 500 mg (one/two/three times per day), to control their diabetes during the period of this study as previously, and acupuncture treatment including electro body acupuncture and Auricular acupuncture for 30 minutes, 10 times, every other day, for 3 weeks.
  metformin
  acupuncture: Electro body acupuncture and auricular acupuncture
- Metformin & Placebo: Metformin 500 mg (one/two/three times per day) to control their diabetes during the period of this study as previously, and placebo acupuncture treatment, needling not in right acupoints and electro acupuncture (EA) machine was switched off during 30 minutes of therapeutic time. And ear acupuncture was just used sticky layers without seeds. All placebo treatments used for 30 minutes, 10 times, every other day, for 3 weeks.
Period: Overall Study
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As a result, 39 participants were distributed by permuted-block randomization. 19 participants were assigned to the case group and 20 to the control group by an independent research assistant, and according to the above-mentioned method of randomization.
Groups:
- Metformin & Acupuncture: Metformin 500 mg, to control their diabetes during the period of this study as previously (with different therapeutic dosage) and acupuncture treatment including electro body acupuncture and Auricular acupuncture for 30 minutes, 10 times, every other day, for 3 weeks.
  metformin
  acupuncture: Electro body acupuncture and auricular acupuncture
- Metformin & Placebo: Metformin 500 mg, to control their diabetes during the period of this study as previously (with different therapeutic dosage) and placebo ( for acupuncture treatment including electro body acupuncture and Auricular acupuncture), needling not in right acupoints (for those points that were located in the abdomen, needles were inserted 0.3 cm laterally from the real location and the needling was maximally superficial. Those points that were located on other parts of the body, needles were inserted 0.5 cm up and 0.5 cm laterally from the real location and needling was superficial as well. Electric lines were connected with some of the needles same way they were connected in another case group. EA machine was switched off during 30 minutes of therapeutic time. Ear acupuncture was used on the same location as in the case group however we just used sticky layers without seeds), for 30 minutes, 10 times, every other day, for 3 weeks.
  metformin Placebo (for acupuncture including electro
- Total: Total of all reporting groups
Arm/Group | Metformin & Acupuncture | Metformin & Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Customized [Mean (Standard Deviation); unit: years] — Patients between 20 and 65 years old of either gender
  years
    Mean age | 42.2 (3.5) | 40.5 (2.6) | 41.3 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: The effect of Metformin and acupuncture combined therapy on weight loss (Change from baseline in body weight), body weight was measured while the subjects were dressed in light clothing after an overnight fasting and by a standard scale to an accuracy of +/-0.1 kg. All measures were recorded by one assessment, at baseline before the first time treatment, and before the last time treatment at week 3.
Time Frame: baseline, week 3
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Metformin & Placebo: Metformin 500 mg (one/two/three times per day), to control their diabetes during the period of this study as previously, and placebo acupuncture treatment, needling not in right acupoints and EA machine was switched off during 30 minutes of therapeutic time. For ear acupuncture was just used sticky layers without seeds. All placebo treatment used for 30 minutes, 10 times, every other day, for 3 weeks.
  metformin
  Placebo acupuncture including placebo EA and auricular acupuncture
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
kg | -4.1 (1.1) | -1.5 (0.3)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

2. Primary Outcome: Fasting Blood Sugar (FBS)
Description: changes FBS, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Metformin & Placebo: Metformin 500 mg (one/two/three times per day), to control their diabetes during the period of this study as previously, and placebo acupuncture treatment, needling not in right acupoints and EA machine was switched off during 30 minutes of therapeutic time. For ear acupuncture was just used sticky layers without seeds. All placebo treatment used for 30 minutes, 10 times, every other day, for 3 weeks.
  metformin
  Placebo EA and auricular acupuncture
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
mmol/L
  FBS blood concentration at the 1th sample, baselin | 6.65 (0.6) | 6.67 (0.5)
  FBS blood concentration at the 2th sample, week 2 | 6.44 (0.5) | 6.55 (0.5)
  FBS blood concentration at the 3th sample, week 3 | 6.12 (0.5) | 6.54 (0.5)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

3. Primary Outcome: Fasting Insulin (FINS)
Description: change of FINS,Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: µIU/ml
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
µIU/ml
  FINS blood level at the 1th sample, baseline | 14.47 (0.8) | 14.45 (0.7)
  FINS blood level at the 2th sample, week 2 | 12.92 (0.7) | 13.75 (0.7)
  FINS blood level at the 3th sample, week 3 | 9.91 (0.7) | 13.6 (0.8)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

4. Primary Outcome: Interleukin-6 (IL-6)
Description: IL-6 changes, IL-6 were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: Pg/dl
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
Pg/dl
  IL-6 blood level at the 1th sample, baseline | 1.44 (0.03) | 1.43 (0.02)
  IL-6 blood level at the 2th sample, week 2 | 1.30 (0.04) | 1.41 (0.02)
  IL-6 blood level at the 3th sample, week 3 | 1.09 (0.05) | 1.37 (0.04)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

5. Primary Outcome: Tumor Necrosis Factor-α (TNF-α)
Description: Blood markers changes in TNF α, were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
Pg/ml
  TNF-α blood level at the 1th sample, baseline | 1.44 (0.02) | 1.44 (0.02)
  TNF-α blood level at the 2th sample, week 2 | 1.42 (0.04) | 1.43 (0.02)
  TNF-α blood level at the 3th sample, week 3 | 1.41 (0.05) | 1.43 (0.02)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p = 0.04, ANOVA

6. Primary Outcome: C-reaction Protein (CRP)
Description: CRP blood markers changes; Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
mg/dl
  CRP blood level at the 1th sample, baseline | 0.60 (0.03) | 0.59 (0.03)
  CRP blood level at the 2th sample, week 2 | 0.59 (0.03) | 0.58 (0.03)
  CRP blood level at the 3th sample, week 3 | 0.57 (0.03) | 0.57 (0.03)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Non-Inferiority or Equivalence — multiple comparatives; p = 0.082, ANOVA — CRP is known to be an independent parameter
Statistical Analysis 2: Comparison: Metformin & Acupuncture; Test type: Non-Inferiority or Equivalence — from 0.60±0.03 mg/dl before treatment to 0.57±0.03 mg/dl after treatment, P=0.082; p = 0.082, ANOVA — CRP is known to be an independent parameter
Statistical Analysis 3: Comparison: Metformin & Placebo; Test type: Non-Inferiority or Equivalence — from 0.59±0.03 mg/dl before treatment to 0.57±0.03 mg/dl after treatment, P=0.082; p = 0.082, ANOVA — CRP is known to be an independent parameter

7. Primary Outcome: Free Fatty Acids (FFAs)
Description: Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
mmol/L
  FFAs blood level at the 1th sample, baseline | 0.72 (0.04) | 0.72 (0.04)
  FFAs blood level at the 2th sample, week 2 | 0.61 (0.03) | 0.70 (0)
  FFAs blood level at the 3th sample, week 3 | 0.51 (0.03) | 0.63 (0.04)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

8. Primary Outcome: Triglyceride (TG)
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
mmol/L
  TG blood level at the 1th sample, baseline | 2.59 (0.6) | 2.69 (0.7)
  TG blood level at the 2th sample, week 2 | 2.44 (0.6) | 2.69 (0.7)
  TG blood level at the 3th sample, week 3 | 2.24 (0.5) | 2.65 (0.7)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

9. Primary Outcome: Low Density Lipoprotein Cholesterol (LDLc)
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
mmol/L
  LDLc blood level at the 1th sample, baseline | 4.05 (0.5) | 4.08 (0.5)
  LDLc blood level at the 2th sample, week 2 | 3.88 (0.5) | 4.0 (0.5)
  LDLc blood level at the 3th sample, week 3 | 3.68 (0.5) | 3.95 (0.5)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

10. Primary Outcome: High Density Lipoprotein Cholesterol (HDLc)
Description: HDLc changes, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
mmol/L
  HDLc blood level at the 1th sample, baseline | 1.08 (0.1) | 1.16 (0.1)
  HDLc blood level at the 2th sample, week 2 | 1.20 (0.1) | 1.21 (0.1)
  HDLc blood level at the 3th sample, week 3 | 1.29 (0.1) | 1.25 (0.1)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

11. Primary Outcome: Ceramides
Description: Changes in ceramides blood level, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
g/dl
  ceramides blood level at the 1th sample, baseline | 8.06 (0.2) | 7.92 (0.2)
  ceramides blood level at the 2th sample, week 2 | 7.24 (0.3) | 7.45 (0.2)
  ceramides blood level at the 3th sample, week 3 | 6.06 (0.3) | 7.18 (0.2)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

12. Primary Outcome: Leptin
Description: changes in Leptin blood level, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
ng/ml
  Leptin blood level at the 1th sample, baseline | 13.32 (0.2) | 13.35 (0.2)
  Leptin blood level at the 2th sample, week 2 | 11.58 (0.4) | 12.67 (0.4)
  Leptin blood level at the 3th sample, week 3 | 10.84 (0.4) | 12.60 (0.4)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

13. Primary Outcome: Adiponectin
Description: Changes in Adiponectin blood level, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
µg/ml
  Adiponectin blood level at the baseline | 7.47 (0.3) | 7.48 (0.2)
  Adiponectin blood level at the 2th sample, week 2 | 8.26 (0.2) | 7.58 (0.3)
  Adiponectin blood level at the 3th sample, week 3 | 8.73 (0.2) | 7.73 (0.3)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

14. Primary Outcome: Glucagon-like Peptide-1 (GLP-1)
Description: changes in GLP-1 blood level, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
mmol/L
  GLP-1 blood level at the 1th sample, baseline | 3.77 (0.2) | 3.75 (0.2)
  GLP-1 blood level at the 2th sample, week 2 | 3.49 (0.2) | 3.50 (0.2)
  GLP-1 blood level at the 3th sample, week 3 | 3.21 (0.1) | 3.43 (0.2)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

15. Primary Outcome: Resistin
Description: Changes in Resistin blood level, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
ng/ml
  Resistin blood level at the 1th sample, baseline | 7.43 (0.2) | 7.36 (0.2)
  Resistin blood level at the 2th sample, week 2 | 6.34 (0.3) | 6.76 (0.2)
  Resistin blood level at the 3th sample, week 3 | 5.24 (0.3) | 6.54 (0.1)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

16. Primary Outcome: Serotonin
Description: changes in Serotonin blood level, Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
ng/ml
  Serotonin blood level at the 1th sample, baseline | 130.4 (3) | 128 (2)
  Serotonin blood level at the 2th sample, week 2 | 144.9 (2) | 135.1 (2)
  Serotonin blood level at the 3th sample, week 3 | 170.5 (3) | 147 (3)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

17. Secondary Outcome: Body Mass Index (BMI)
Description: change of BMI. Body height was measured to an accuracy of +/-0.1cm. BMI was calculated by dividing weight (kg) into height (squared m²).
Time Frame: baseline, week 3
Measure: Mean (Standard Deviation); unit: Kg/m²
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
Kg/m²
  BMI blood level at the 1th sample, baseline | 27.6 (2.5) | 28.2 (1.6)
  BMI blood level at the 3th sample, week 3 | 26.2 (2.4) | 27.7 (1.6)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

18. Secondary Outcome: HOMA-IR
Description: Changes of IR was calculated by the homeostasis model (HOMA-IR), proposed by Matthews et al. HOMA-IR = (fasting insulin (mmol/L) × fasting glucose (µIU/ml))/22•5. Blood markers were calculated by measuring them after drawing 10 ml of blood from cubital vein in each patient, after 8 hours of overnight fasting and before treatment; Blood was collected three times during the study (at the beginning, at the 5th time, and at the end), from groups, using standard range and ELISA diagnostic kits (Biomatik USA LLC, www.biomatik.com), and clinical assessments and measurements undertaken after 3 weeks. Readings/assessment was performed at 3 weeks.
Time Frame: baseline, week 2, week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Number analyzed (Participants) | 19 | 20
units on a scale
  HOMA-IR at the 1th sample, baseline | 4.25 (0.2) | 4.36 (0.6)
  HOMA-IR at the 2th sample, week 2 | 3.68 (0.1) | 4.06 (0.5)
  HOMA-IR at the 3th sample, week 3 | 2.67 (0.1) | 4.01 (0.5)
Statistical Analysis 1: Comparison: Metformin & Acupuncture vs Metformin & Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: 3 WEEKS
Description: All participants were treated 10 times every other day, for a total duration of 3 weeks.
Arm/Group | Metformin & Acupuncture | Metformin & Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No